CLINICAL TRIAL: NCT03697018
Title: Evaluation of Antagonist Wear Behavior and Patient Satisfaction of Monolithic Zirconia Versus Lithium Silicate Zirconia Crowns
Brief Title: Evaluation of Antagonist Wear Behavior and Patient Satisfaction of Zirconia Reinforced Lithium Silicate Glass When Compared to Monolithic Zirconia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Hany, PHD candidate, fixed prosthodontic department, faculty of Oral and dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-10-01
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Wear of the Natural Enamel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zirconia reinforced lithium silicate glass ceramic (Experimental): It represent a new generation of glass ceramic material, enriched with zirconia (10% by weight), the material offers natural esthetics with successful outcome.
  Interventions: Other: zirconia reinforced lithium silicate glass ceramic
- monolithic zirconia (Active Comparator): Zirconia or zirconium dioxide (ZrO2) is a highly attractive ceramic material in prosthodontics due to its excellent mechanical properties. It is widely used to build prosthetic devices.
  Interventions: Other: zirconia reinforced lithium silicate glass ceramic

INTERVENTIONS:
Other: zirconia reinforced lithium silicate glass ceramic — It represent a new generation of glass ceramic material. Using an innovative manufacturing process the glass ceramic is enriched with zirconia (10% by weight) for dental CAD/CAM applications for the fabrication of inlays, onlays, crowns and anterior and posterior single tooth restorations on implant abutments.

SUMMARY:
evaluation of wear behavior and patient satisfaction of monolithic zirconia and zirconia reinforced glass crowns after follow-up periods 0,3,6,12 months.

DETAILED DESCRIPTION:
two groups of patients will be selected according to special inclusion criteria n=13 in each group total of 26. each group will receive one of the crowns used in this study either ( monolithic zirconia or zirconia reinforced lithium silicate glass) after crown delivery wear and patient satisfaction will be recorded at 0,3,6,12 moths follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age range from 20-60 to be able to read and write in order to sign the informed consent document.
2. Patients physically and psychologically able to tolerate conventional restorative procedures.
3. Patients with no active periodontal and or pulpal diseases, having teeth with good restorations.
4. Patients with root canal treated teeth requiring full coverage restorations.
5. Patients indicated for full coverage (e.g. moderate to severe discoloration, coronal fracture, malposed or malformed teeth).
6. Patients willing to return for follow-up examinations and assessments

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patient with poor oral hygiene.
3. Patients with psychiatric problems or unrealistic expectations
4. Patient with no opposite occluding dentition in the area intended for restoration.
5. Patient suffering from Para functional habits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
wear of the antagonist natural enamel | from baseline till one year
  loss of opposing tooth structure which will be measured by 3D Profilometer

SECONDARY OUTCOMES:
patient satisfaction | from baseline till one year
  visual analogue scale (VAS): scale range from 0-10 for describing the intensity of pain the patient suffering. 0: no pain, 5: moderate pain, 10: unbearable pain.

IPD SHARING:
Plan to Share IPD: Undecided
conditions and factors which increase degree and progression of wear and clinical behavior of monolithic zirconia and zirconia reinforced lithium silicate restorations.